CLINICAL TRIAL: NCT03538743
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO ASSESS THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF MULTIPLE ESCALATING ORAL DOSES OF PF-06882961 IN ADULT SUBJECTS WITH TYPE 2 DIABETES MELLITUS
Brief Title: 4-Week, Multiple-dose, Dose-escalating Study In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C3421002
Record Dates: First submitted 2018-05-07; First posted 2018-05-29 (Actual); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06882961 30 mg (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 100 mg (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 300 mg (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 600 mg (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 dose TBD Cohort 5 (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 dose TBD Cohort 6 (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 dose TBD Cohort 7 (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 dose TBD Cohort 8 (Experimental)
  Interventions: Drug: PF-06882961

INTERVENTIONS:
Drug: Placebo — Tablet, 0 mg, twice daily, 28 days
  Arms: Placebo
Drug: PF-06882961 — Tablet, 15 mg twice daily, 28 days
  Arms: PF-06882961 30 mg
Drug: PF-06882961 — Tablet, 50 mg twice daily, 28 days
  Arms: PF-06882961 100 mg
Drug: PF-06882961 — Tablet, 150 mg twice daily, 28 days
  Arms: PF-06882961 300 mg
Drug: PF-06882961 — Tablet, 300 mg twice daily, 28 days
  Arms: PF-06882961 600 mg
Drug: PF-06882961 — Tablet, dose TBD, twice daily, Cohort 5, 28 days
  Arms: PF-06882961 dose TBD Cohort 5
Drug: PF-06882961 — Tablet, dose TBD, twice daily, Cohort 6, 28 days
  Arms: PF-06882961 dose TBD Cohort 6
Drug: PF-06882961 — Tablet, dose TBD, twice daily, Cohort 7, 28 days
  Arms: PF-06882961 dose TBD Cohort 7
Drug: PF-06882961 — Tablet, dose TBD, twice daily, Cohort 8, 28 days
  Arms: PF-06882961 dose TBD Cohort 8

SUMMARY:
This is a dose-escalating study in patients with Type 2 diabetes on metformin. Participants will receive an investigational product or placebo for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with a stable dose of metformin at least 500 mg
* HbA1c value between 7.0 and 10.5%

Exclusion Criteria:

- Type 1 diabetes or secondary forms of diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Qps-Mra, Llc, South Miami, Florida
  - Qps-Mra,Llc, South Miami, Florida
  - Altasciences Clinical Kansas, Inc., Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Saxena AR, Gorman DN, Esquejo RM, Bergman A, Chidsey K, Buckeridge C, Griffith DA, Kim AM. Danuglipron (PF-06882961) in type 2 diabetes: a randomized, placebo-controlled, multiple ascending-dose phase 1 trial. Nat Med. 2021 Jun;27(6):1079-1087. doi: 10.1038/s41591-021-01391-w. Epub 2021 Jun 14. PMID 34127852
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421002

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-06882961 was administered orally once daily (QD) or twice daily (BID) (dependent upon corresponding study treatment regimen) for a total of 28 days.
- PF-06882961 10mg BID: PF-06882961 tablet was administered orally at 5 mg BID from Day 1 to Day 14 followed by a dose of 10 mg BID from Day 15 to Day 28.
- PF-06882961 15mg BID: PF-06882961 tablet was administered orally at 15 mg BID for a total of 28 days.
- PF-06882961 50mg BID: PF-06882961 tablet was administered orally at 50 mg BID for a total of 28 days.
- PF-06882961 70mg BID: PF-06882961 tablet was administered orally at 20 mg (Day 1-3), 40 mg (Day 4-6), 50 mg (Day 7-9) and 70 mg (Day 10-28) BID for a total of 28 days.
- PF-06882961 120mg BID: PF-06882961 tablet was administered orally at 20 mg (Day 1-2), 40 mg (Day 3-4), 60 mg (Day 5-6), 80 mg (Day 7-9), 100 mg (Day 10-12) and 120 mg (Day 13-28) BID for a total of 28 days.
- PF-06882961 120mg BID Slow Titration (ST): PF-06882961 tablet was administered orally at 10 mg (Day 1-4), 20 mg (Day 5-8), 40 mg (Day 9-12), 60 mg (Day 13-16), 80 mg (Day 17-20), 100 mg (Day 21-24) and 120 mg (Day 25-28) BID for a total of 28 days.
- PF-06882961 120mg QD: PF-06882961 tablet was administered orally at 10 mg (Day 1-2), 20 mg (Day 3-4), 30 mg (Day 5-6), 40 mg (Day 7-10), 60 mg (Day 11-14), 80 mg (Day 15-18), 100 mg (Day 19-22) and 120 mg (Day 23-28) QD for a total of 28 days.
- PF-06882961 200mg QD Controlled Release (CR): PF-06882961 CR tablet was administered orally at 50 mg (Day 1-7), 100 mg (Day 8-14), 150 mg (Day 15-21) and 200 mg (Day 22-28) QD for a total of 28 days.
Period: Overall Study
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID Slow Titration (ST) | PF-06882961 120mg QD | PF-06882961 200mg QD Controlled Release (CR)
Started | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10
Received Treatment | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10
Completed | 25 | 9 | 8 | 8 | 9 | 9 | 9 | 8 | 7
Not Completed | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Treatment-Related Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Groups:
- Placebo: Placebo matched to PF-06882961 was administered orally QD or BID(dependent upon corresponding study treatment regimen) for a total of 28 days.
- PF-06882961 120mg BID ST: PF-06882961 tablet was administered orally at 10 mg (Day 1-4), 20 mg (Day 5-8), 40 mg (Day 9-12), 60 mg (Day 13-16), 80 mg (Day 17-20), 100 mg (Day 21-24) and 120 mg (Day 25-28) BID for a total of 28 days.
- PF-06882961 200mg QD CR: PF-06882961 CR tablet was administered orally at 50 mg (Day 1-7), 100 mg (Day 8-14), 150 mg (Day 15-21) and 200 mg (Day 22-28) QD for a total of 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID ST | PF-06882961 120mg QD | PF-06882961 200mg QD CR | Total
Number analyzed (Participants) | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10 | 98
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  45-64 years | 19 | 8 | 6 | 6 | 8 | 8 | 7 | 7 | 8 | 77
  >=65 years | 5 | 0 | 2 | 4 | 1 | 0 | 2 | 1 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 6 | 5 | 5 | 2 | 5 | 4 | 5 | 47
  Male | 12 | 7 | 3 | 5 | 4 | 7 | 4 | 4 | 5 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 6 | 4 | 7 | 6 | 4 | 4 | 6 | 6 | 61
  Not Hispanic or Latino | 7 | 3 | 5 | 3 | 3 | 5 | 5 | 2 | 4 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 7 | 5 | 8 | 7 | 6 | 4 | 8 | 7 | 70
  Black or African American | 7 | 2 | 3 | 2 | 2 | 3 | 5 | 0 | 3 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Age Range [Median (Full Range); unit: Years] | 60.0 [41 to 70] | 55.0 [44 to 61] | 55.0 [37 to 68] | 63.5 [48 to 68] | 60.0 [46 to 65] | 57.0 [40 to 64] | 58.0 [50 to 69] | 58.0 [53 to 66] | 59.0 [45 to 69] | 58.0 [37 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-causality and Treatment-related Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-related adverse event (AE) was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Any such events with initial onset or increasing in severity after the first dose of study treatment were counted as treatment-emergent.
Time Frame: From baseline to up to 35 days after last dose for a total of approximately 63 days
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID ST | PF-06882961 120mg QD | PF-06882961 200mg QD CR
Number analyzed (Participants) | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10
Participants
  All-causality AE | 17 | 6 | 8 | 10 | 8 | 8 | 9 | 8 | 9
  All-causality SAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Treatment-related AE | 14 | 4 | 4 | 10 | 7 | 8 | 9 | 8 | 9
  Treatment-related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology (hemoglobin, hematocrit, erythrocytes, reticulocytes, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time, prothrombin time [PT], PT/international normalized ratio, reticulocytes); chemistry (indirect bilirubin, direct bilirubin, protein, albumin, blood urea nitrogen, creatinine, creatine kinase, urate, calcium, sodium, potassium, chloride, bicarbonate, urine urobilinogen); urinalysis (pH, urine glucose, urine ketones, urine protein, urine hemoglobin, nitrites, leukocyte esterase, urine erythrocytes, urine leukocytes, urine hyaline casts, urine bilirubin).
Time Frame: From baseline to up to 14 days after last dose for a total of approximately 42 days
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID ST | PF-06882961 120mg QD | PF-06882961 200mg QD CR
Number analyzed (Participants) | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10
Participants | 24 | 7 | 8 | 10 | 8 | 8 | 9 | 7 | 10

3. Primary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs categorical summarization criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine SBP greater than or equal to (>=) 30 mmHg; 5) change from baseline (increase or decrease) in supine DBP >= 20 mmHg.
Time Frame: From baseline to up to 14 days after last dose for a total of approximately 42 days
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID ST | PF-06882961 120mg QD | PF-06882961 200mg QD CR
Number analyzed (Participants) | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10
Participants
  Supine SBP <90 mmHg | 3 | 3 | 2 | 1 | 3 | 0 | 3 | 0 | 1
  Supine SBP increase >=30 mmHg | 4 | 0 | 0 | 2 | 3 | 1 | 2 | 2 | 1
  Supine SBP decrease >=30 mmHg | 9 | 2 | 5 | 3 | 5 | 3 | 3 | 5 | 4
  Supine DBP <50 mmHg | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 0
  Supine DBP increase >=20 mmHg | 1 | 1 | 1 | 0 | 4 | 1 | 2 | 2 | 1
  Supine DBP decrease >=20 mmHg | 6 | 2 | 1 | 2 | 1 | 3 | 4 | 2 | 3
  Supine pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Interval
Description: ECG categorical summarization criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) greater than or equal to (>=) 300 millisecond (msec), b) >=25% increase when baseline is > 200 msec or >=50% increase when baseline is less than or equal to (<=) 200 msec.
  2. QRS duration (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) >=140 msec, b) >=50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and <=480 msec, b) >480 msec and <=500 msec, c) >500 msec, d) >30 msec and <=60 msec increase from baseline, e) >60 msec increase from baseline
Time Frame: From baseline to up to 14 days after last dose for a total of approximately 42 days
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID ST | PF-06882961 120mg QD | PF-06882961 200mg QD CR
Number analyzed (Participants) | 25 | 9 | 9 | 10 | 9 | 9 | 9 | 8 | 10
Participants
  PR interval ≥300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in PR interval ≥25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration ≥140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in QRS duration ≥50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >450 and ≤480 msec | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >480 and ≤500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in QTcF interval >30 and ≤60 msec | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Change in QTcF interval >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: AUC24 and AUCtau of PF-06882961 on Day 1, Day 14 or 21 and Day 28
Description: Area under the concentration-time profile from time zero to time 24 hours (AUC24) was calculated as AUCtau1 +AUCtau2, where AUCtau was area under the plasma concentration-time profile from time zero to time tau (tau1 = 0 to 10 hours and tau2=10 to 24 hours). AUCtau was determined using linear/log trapezoidal method.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 14 and 24 hrs post dose on Day 1, 14 or 21, and 28
Population: All randomized participants who received at least 1 dose of PF-06882961 and who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram.hours/milliliter (ng.h/mL)
Groups:
- PF-06882961 15mg BID (Cohort 1): PF-06882961 tablet was administered orally at 15 mg BID for a total of 28 days.
- PF-06882961 50mg BID (Cohort 2): PF-06882961 tablet was administered orally at 50 mg BID for a total of 28 days.
- PF-06882961 70mg BID (Cohort 3): PF-06882961 tablet was administered orally at 20 mg (Day 1-3), 40 mg (Day 4-6), 50 mg (Day 7-9) and 70 mg (Day 10-28) BID for a total of 28 days.
- PF-06882961 120mg BID (Cohort 4): PF-06882961 tablet was administered orally at 20 mg (Day 1-2), 40 mg (Day 3-4), 60 mg (Day 5-6), 80 mg (Day 7-9), 100 mg (Day 10-12) and 120 mg (Day 13-28) BID for a total of 28 days.
- PF-06882961 10mg BID (Cohort 5): PF-06882961 tablet was administered orally at 5 mg BID from Day 1 to Day 14 followed by a dose of 10 mg BID from Day 15 to Day 28.
- PF-06882961 120mg BID ST (Cohort 6): PF-06882961 tablet was administered orally at 10 mg (Day 1-4), 20 mg (Day 5-8), 40 mg (Day 9-12), 60 mg (Day 13-16), 80 mg (Day 17-20), 100 mg (Day 21-24) and 120 mg (Day 25-28) BID for a total of 28 days.
- PF-06882961 200mg QD CR (Cohort 7): PF-06882961 CR tablet was administered orally at 50 mg (Day 1-7), 100 mg (Day 8-14), 150 mg (Day 15-21) and 200 mg (Day 22-28) QD for a total of 28 days.
- PF-06882961 120mg QD (Cohort 8): PF-06882961 tablet was administered orally at 10 mg (Day 1-2), 20 mg (Day 3-4), 30 mg (Day 5-6), 40 mg (Day 7-10), 60 mg (Day 11-14), 80 mg (Day 15-18), 100 mg (Day 19-22) and 120 mg (Day 23-28) QD for a total of 28 days.
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 9 | 9 | 10 | 8
nanogram.hours/milliliter (ng.h/mL)
  AUC24 on Day 1 | 707.5 (43) | 1502 (29) | 645.8 (52) | 666.1 (54) | 178.7 (72) | 324.0 (41) | 393.9 (80) | 184.6 (49)
  AUCtau1 on Day 1 | 288.1 (37) | 741.4 (35) | 279.7 (49) | 260.3 (45) | 74.50 (66) | 147.7 (43) | NA (NA) — Data was calculated as AUC24 only for QD dosing. | NA (NA) — Data was calculated as AUC24 only for QD dosing.
  AUCtau2 on Day 1 | 414.8 (50) | 678.5 (79) | 364.9 (56) | 401.9 (62) | 103.7 (76) | 176.4 (42) | NA (NA) — Data was calculated as AUC24 only for QD dosing. | NA (NA) — Data was calculated as AUC24 only for QD dosing.
  AUC24 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  AUC24 on Day 14 or 21 | 853.8 (45) | 2092 (91) | 2988 (59) | 8149 (84) | 201.6 (63) | 2660 (76) | 1291 (68) | 1204 (43)
  AUCtau1 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  AUCtau1 on Day 14 or 21 | 348.6 (48) | 880.3 (78) | 1462 (70) | 3772 (85) | 85.57 (59) | 957.3 (66) | NA (NA) — Data was calculated as AUC24 only for QD dosing. | NA (NA) — Data was calculated as AUC24 only for QD dosing.
  AUCtau2 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  AUCtau2 on Day 14 or 21 | 500.1 (46) | 1175 (110) | 1517 (53) | 4361 (89) | 115.4 (68) | 1693 (83) | NA (NA) — Data was calculated as AUC24 only for QD dosing. | NA (NA) — Data was calculated as AUC24 only for QD dosing.
  AUC24 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 7
  AUC24 on Day 28 | 876.7 (41) | 1653 (55) | 3171 (56) | 8368 (79) | 455.9 (66) | 5973 (87) | 4372 (31) | 2723 (39)
  AUCtau1 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 8
  AUCtau1 on Day 28 | 331.1 (40) | 671.1 (35) | 1153 (44) | 3534 (87) | 190.8 (60) | 2249 (88) | NA (NA) — Data was calculated as AUC24 only for QD dosing. | NA (NA) — Data was calculated as AUC24 only for QD dosing.
  AUCtau2 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 8
  AUCtau2 on Day 28 | 534.7 (46) | 960.1 (73) | 1970 (68) | 4852 (74) | 261.0 (72) | 3668 (91) | NA (NA) — Data was calculated as AUC24 only for QD dosing. | NA (NA) — Data was calculated as AUC24 only for QD dosing.

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-06882961 on Day 1, Day 14 or 21 and Day 28
Description: For BID dosing, parameters were calculated for both dosing intervals (0-10 hr = interval 1 and 10-24 hr = interval 2) and were displayed as Cmax1, Cmax2.
  Cmax1: maximum plasma concentration during the dosing interval τ1 =0 to 10 hours.
  Cmax2: maximum plasma concentration during the dosing interval τ2=10 to 24 hours.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 14 and 24 hours post dose on Day 1, 14 or 21, and 28
Population: All randomized participants treated who had at least 1 measurable concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 9 | 9 | 10 | 8
nanogram/milliliter (ng/mL)
  Cmax on Day 1 | 50.58 (40) | 124.4 (51) | 49.75 (50) | 51.61 (50) | 15.02 (70) | 26.02 (39) | 28.67 (87) | 20.40 (29)
  Cmax1 on Day 1 | 42.69 (29) | 119.1 (56) | 45.01 (48) | 36.51 (43) | 12.82 (58) | 24.06 (42) | NA (NA) — Data was calculated as Cmax only for QD dosing. | NA (NA) — Data was calculated as Cmax only for QD dosing.
  Cmax2 on Day 1 | 40.63 (66) | 68.77 (51) | 42.33 (59) | 44.97 (61) | 13.98 (75) | 21.64 (41) | NA (NA) — Data was calculated as Cmax only for QD dosing. | NA (NA) — Data was calculated as Cmax only for QD dosing.
  Cmax on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  Cmax on Day 14 or 21 | 65.78 (35) | 149.8 (88) | 253.6 (76) | 788.4 (89) | 18.63 (47) | 188.5 (57) | 98.11 (54) | 100.7 (35)
  Cmax1 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  Cmax1 on Day 14 or 21 | 55.00 (43) | 130.2 (85) | 235.1 (84) | 682.7 (92) | 15.31 (50) | 143.0 (71) | NA (NA) — Data was calculated as Cmax only for QD dosing. | NA (NA) — Data was calculated as Cmax only for QD dosing.
  Cmax2 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  Cmax2 on Day 14 or 21 | 63.89 (36) | 127.9 (86) | 202.8 (50) | 505.3 (93) | 17.16 (58) | 178.4 (56) | NA (NA) — Data was calculated as Cmax only for QD dosing. | NA (NA) — Data was calculated as Cmax only for QD dosing.
  Cmax on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 7
  Cmax on Day 28 | 81.56 (32) | 133.7 (69) | 328.8 (49) | 685.2 (87) | 38.38 (58) | 437.6 (94) | 303.9 (32) | 192.2 (52)
  Cmax1 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 8
  Cmax1 on Day 28 | 50.24 (44) | 103.8 (50) | 197.9 (51) | 649.2 (90) | 30.42 (52) | 357.1 (84) | NA (NA) — Data was calculated as Cmax only for QD dosing. | NA (NA) — Data was calculated as Cmax only for QD dosing.
  Cmax2 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 8
  Cmax2 on Day 28 | 74.22 (37) | 117.2 (63) | 306.5 (49) | 617.9 (93) | 35.01 (56) | 410.3 (90) | NA (NA) — Data was calculated as Cmax only for QD dosing. | NA (NA) — Data was calculated as Cmax only for QD dosing.

7. Secondary Outcome: Time for Cmax (Tmax) of PF-06882961 on Day 1, Day 14 or 21 and Day 28
Description: Time for Cmax, Cmax1 and Cmax2 (Tmax, Tmax1 and Tmax2) of PF-06293620 was observed directly from data as time of first occurrence.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 14 and 24 hrs post dose on Day 1, 14 or 21, and 28
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 9 | 9 | 10 | 8
hours
  Tmax on Day 1 | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | 13.0 [8.00 to 23.9] | 3.00 [1.00 to 6.00]
  Tmax1 on Day 1 | 4.00 [2.00 to 8.00] | 4.00 [1.00 to 6.00] | 2.00 [1.00 to 6.00] | 4.00 [2.00 to 6.00] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | NA [NA to NA] — Data was calculated as Tmax only for QD dosing. | NA [NA to NA] — Data was calculated as Tmax only for QD dosing.
  Tmax2 on Day 1 | 14.0 [10.0 to 24.0] | 14.0 [10.0 to 24.0] | 14.0 [12.0 to 14.0] | 14.0 [12.0 to 24.0] | 12.0 [12.0 to 14.0] | 14.0 [12.0 to 24.0] | NA [NA to NA] — Data was calculated as Tmax only for QD dosing. | NA [NA to NA] — Data was calculated as Tmax only for QD dosing.
  Tmax on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  Tmax on Day 14 or 21 | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | 12.0 [6.00 to 14.0] | 6.00 [4.00 to 10.0]
  Tmax1 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  Tmax1 on Day 14 or 21 | 4.00 [2.00 to 8.00] | 4.00 [1.00 to 6.00] | 1.05 [1.00 to 6.00] | 1.54 [1.00 to 6.00] | 6.00 [1.00 to 6.00] | 6.00 [4.00 to 10.0] | NA [NA to NA] — Data was calculated as Tmax only for QD dosing. | NA [NA to NA] — Data was calculated as Tmax only for QD dosing.
  Tmax2 on Day 14 or 21: number analyzed (Participants) | 8 | 4 | 9 | 8 | 9 | 9 | 10 | 8
  Tmax2 on Day 14 or 21 | 13.0 [12.0 to 14.0] | 13.0 [10.0 to 14.0] | 12.0 [12.0 to 12.0] | 12.0 [10.0 to 14.0] | 12.0 [12.0 to 14.0] | 14.0 [12.0 to 24.0] | NA [NA to NA] — Data was calculated as Tmax only for QD dosing. | NA [NA to NA] — Data was calculated as Tmax only for QD dosing.
  Tmax on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 7
  Tmax on Day 28 | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | NA [NA to NA] — Data was calculated as Tmax1 and Tmax2 only for BID dosing. | 14.0 [8.00 to 14.0] | 10.0 [6.00 to 14.0]
  Tmax1 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 7
  Tmax1 on Day 28 | 5.00 [4.00 to 8.00] | 3.00 [0.00 to 8.00] | 6.00 [2.00 to 8.00] | 4.00 [1.00 to 6.00] | 4.00 [2.00 to 8.00] | 6.00 [4.00 to 10.0] | NA [NA to NA] — Data was calculated as Tmax only for QD dosing. | NA [NA to NA] — Data was calculated as Tmax only for QD dosing.
  Tmax2 on Day 28: number analyzed (Participants) | 8 | 4 | 8 | 8 | 9 | 7 | 7 | 7
  Tmax2 on Day 28 | 12.0 [12.0 to 14.0] | 12.0 [12.0 to 12.0] | 12.0 [12.0 to 14.0] | 12.0 [12.0 to 14.0] | 12.0 [12.0 to 14.0] | 12.0 [10.0 to 14.0] | NA [NA to NA] — Data was calculated as Tmax only for QD dosing. | NA [NA to NA] — Data was calculated as Tmax only for QD dosing.

8. Secondary Outcome: Terminal Half-life (t½) of PF-06882961 on Day 28
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 14 and 24 hrs post dose on Day 28
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 9 | 9 | 10 | 8
hours | 5.100 (1.2186) | 5.067 (0.75593) | 4.681 (0.59504) | 6.203 (2.3505) | 8.090 (3.3234) | 6.730 (2.5056) | 5.773 (1.4876) | 4.954 (0.58819)

9. Secondary Outcome: Amount of Unchanged Drug Recovered in Urine Over 24 Hours (Ae24) of PF-06882961 on Day 28
Description: Ae was the cumulative amount of drug recovered unchanged in urine during the dosing interval, where the dosing interval was 24 hours. Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval. Sample volume = (urine weight in gram [g]/1.020), where 1.020 g/mL was the approximate specific gravity of urine.
Time Frame: 0 to 24 hours post-dose on Day 28
Population: All randomized participants who received at least 1 dose of PF-06882961 and who have at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 8 | 9 | 7 | 7 | 8
microgram | 17.25 (36) | 33.60 (69) | 41.16 (243) | NA (NA) — "NA" indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 14.97 (67) | 62.63 (439) | 72.98 (38) | 49.09 (97)

10. Secondary Outcome: Ae24 (%) of PF-06882961 on Day 28
Description: Percent of dose recovered in urine as unchanged drug. Ae24% = 100* Ae24/Dose
Time Frame: 0 to 24 hours post-dose on Day 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 8 | 9 | 7 | 7 | 8
Percentage | 0.05747 (36) | 0.03360 (69) | 0.02942 (242) | NA (NA) — "NA" indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.07483 (67) | 0.02607 (439) | 0.03652 (38) | 0.04094 (97)

11. Secondary Outcome: Renal Clearance (CLr) of PF-06882961 on Day 28
Description: CLr was calculated as Ae divided by AUCtau, where dosing interval is 24 hours.
Time Frame: 0 to 24 hours post-dose on Day 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | PF-06882961 15mg BID (Cohort 1) | PF-06882961 50mg BID (Cohort 2) | PF-06882961 70mg BID (Cohort 3) | PF-06882961 120mg BID (Cohort 4) | PF-06882961 10mg BID (Cohort 5) | PF-06882961 120mg BID ST (Cohort 6) | PF-06882961 200mg QD CR (Cohort 7) | PF-06882961 120mg QD (Cohort 8)
Number analyzed (Participants) | 9 | 10 | 9 | 8 | 9 | 7 | 7 | 8
mL/min | 0.3273 (18) | 0.3385 (18) | 0.3094 (70) | NA (NA) — "NA" indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.5470 (26) | 0.2006 (228) | 0.2895 (21) | 0.3178 (73)

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days after last dose for a total of approximately 63 days
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | PF-06882961 10mg BID | PF-06882961 15mg BID | PF-06882961 50mg BID | PF-06882961 70mg BID | PF-06882961 120mg BID | PF-06882961 120mg BID ST | PF-06882961 120mg QD | PF-06882961 200mg QD CR
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/9 | 0/9 | 0/10 | 0/9 | 0/9 | 0/9 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/9 | 0/9 | 0/10 | 0/9 | 0/9 | 1/9 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 15/25 | 6/9 | 8/9 | 10/10 | 8/9 | 8/9 | 9/9 | 8/8 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | PF-06882961 10mg BID (N=9) | PF-06882961 15mg BID (N=9) | PF-06882961 50mg BID (N=10) | PF-06882961 70mg BID (N=9) | PF-06882961 120mg BID (N=9) | PF-06882961 120mg BID ST (N=9) | PF-06882961 120mg QD (N=8) | PF-06882961 200mg QD CR (N=10)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — This event occurred in the follow up period and was assessed as not treatment-related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=25) | PF-06882961 10mg BID (N=9) | PF-06882961 15mg BID (N=9) | PF-06882961 50mg BID (N=10) | PF-06882961 70mg BID (N=9) | PF-06882961 120mg BID (N=9) | PF-06882961 120mg BID ST (N=9) | PF-06882961 120mg QD (N=8) | PF-06882961 200mg QD CR (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 2 | 1 | 0 | 5 | 1 | 0 | 2 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 2 | 1 | 6 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 3 | 2 | 3 | 4 | 1 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 0 | 5 | 4 | 4 | 7 | 3 | 5
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0/0 | 0/0 | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 7 | 3 | 8 | 9 | 7 | 8
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 2 | 7 | 7 | 3 | 3
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroid function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 6 | 2 | 3 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 1
Headache (Nervous system disorders) | 8 | 0 | 1 | 5 | 2 | 0 | 0 | 4 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03538743/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03538743/SAP_001.pdf